CLINICAL TRIAL: NCT02074540
Title: The Influence of Health Beliefs and Uncertainty on Diabetes Type II Patient Compliance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0005-14
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetes Type II Patients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire that is based on socio-demographic characteristics, Morisky's Four-Item Self-Reported Adherence Measure, Becker's Theory of Health Beliefs and Mishel's Theory of Uncertainty

SUMMARY:
To determine the predicting factors and indicators of compliance with insulin treatment in Diabetes Type II patients.

ELIGIBILITY:
Inclusion Criteria:

* With complete cognitive abilities
* Independent functioning
* Take insulin

Exclusion Criteria:

* Critically ill patients
* Psychiatric patients

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes Type II patients who receive insulin and are hospitalized in the Hillel Yaffe Medical Center in a variety of departments. Patients are both Hebrew and Arabic speaking.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Insulin adherence | Forty minutes
  Average number of positive responses on the questionnaire scale

CONTACTS AND LOCATIONS:
Overall Officials: Jalal Ashkar, MD, Study Director — Hillel Yaffe Medical Center; Rinat Majadly, RN, BA, Principal Investigator — Hillel Yaffe Medical Center